CLINICAL TRIAL: NCT04243759
Title: A Smartphone App to Capture Inhibitory Control as a Novel Moderate Drinking Tool for Young Adults
Brief Title: Inhibitory Control Smartphone App
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB202001530; R21AA026918 (NIH); IRB201801604 - N (Other: UF IRB)
Record Dates: First submitted 2020-01-21; First posted 2020-01-28 (Actual); Results first posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2024-12

CONDITIONS: Drinking, Alcohol; Drinking Behavior
MeSH Terms: conditions — Alcohol Drinking; Drinking Behavior

STUDY DESIGN:
Intervention Model Description: Heavy drinking young adults will be randomized to 1 of the 3 apps. After initial use of their randomized app, they will then be dosed to .06% blood alcohol content (BAC) in a naturalistic lab, followed by app use. For 4 weeks post-session, all participants will use the experimental app for 2 weeks in real drinking occasions and not use it the other 2 weeks.
Who Masked: Participant, Care Provider
Masking Description: Staff working with participants will not know app assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control App Group (Experimental): Young Adult Drinkers will be randomized to 1 of the 3 app conditions (Control App Version; Standard App Version; Experimental, Feedback App Version). The apps will be tested both during a laboratory alcohol drinking session and a 4-week period outside the lab in which they can use this technology in actual drinking situations. For the 4-week period outside the lab, all participants will use the experimental app for 2 weeks in real drinking occasions and not use it the other 2 weeks.
  Interventions: Behavioral: Control App Version; Behavioral: Experimental, Feedback App Version
- Standard App Group (Experimental): Young Adult Drinkers will be randomized to 1 of the 3 app conditions (Control App Version; Standard App Version; Experimental, Feedback App Version). The apps will be tested both during a laboratory alcohol drinking session and a 4-week period outside the lab in which they can use this technology in actual drinking situations. For the 4-week period outside the lab, all participants will use the experimental app for 2 weeks in real drinking occasions and not use it the other 2 weeks.
  Interventions: Behavioral: Standard App Version; Behavioral: Experimental, Feedback App Version
- Experimental, Feedback App Group (Experimental): Young Adult Drinkers will be randomized to 1 of the 3 app conditions (Control App Version; Standard App Version; Experimental, Feedback App Version). The apps will be tested both during a laboratory alcohol drinking session and a 4-week period outside the lab in which they can use this technology in actual drinking situations. For the 4-week period outside the lab, all participants will use the experimental app for 2 weeks in real drinking occasions and not use it the other 2 weeks.
  Interventions: Behavioral: Experimental, Feedback App Version

INTERVENTIONS:
Behavioral: Control App Version — The control version is a smartphone-compatible CGNG. The cued go/no-go (CGNG) tests ability to respond fast to "go" targets (activation) while withholding response to "no-go" targets (inhibition).
  Arms: Control App Group
Behavioral: Standard App Version — The standard version is the same as the control version with the exception that information about performance (correct or incorrect) is displayed along with RT in ms for a correct response during each inter-trial interval.
  Arms: Standard App Group
Behavioral: Experimental, Feedback App Version — The experimental, feedback version includes the standard plus feedback on RT and inhibition errors compared to pre-drinking. The app will state that there are simple alternatives with invitation to press a box to view advice, based on research that risk information may increase risky behavior if convenient options are not given73. Feedback will be worded non-judgmentally per motivational interviewing tenets.

SUMMARY:
The proposed study will address a critical knowledge gap: there are no evidence-based smartphone apps for reducing young adult drinking. The purpose of the study is to test alcohol-related smartphone applications designed to provide assistance during actual drinking situations to help young adults reduce their drinking. It is the researchers hypothesis that participants will self-administer less alcohol when using the experimental app with feedback.

DETAILED DESCRIPTION:
An app giving in-the-moment feedback could increase perceived impairment, and reduce drinking and consequences.

The cued go/no-go (CGNG) task is an ideal choice for in-the-moment impairment feedback. Its instructions are simple; practice effects are minimal; and is sensitive to alcohol. The CGNG tests ability to respond fast to "go" targets (activation) while withholding response to "no-go" targets (inhibition). Activation/inhibition tension is externally valid. Dual process models posit risk behaviors stem from overactive appetitive drives that are compelling and hard to inhibit. Poor CGNG performance post-alcohol has been related to poor simulated driving, enhancing external validity. Moderate dosing to .05-.06% blood alcohol content (BAC) reliably increases inhibition errors, but slowing reaction time (RT) to "go" cues requires higher doses. RT to go cues often recovers later in a drinking episode (acute tolerance) but ability to inhibit does not. Thus at this BAC, ability to respond remains but inhibition is impaired, which relates to risk behaviors like DUI as young adults underrate impairment.

ELIGIBILITY:
Inclusion Criteria:

* Be able to read English and complete study evaluations
* Report drinking to an estimated blood alcohol concentration (eBAC) of 0.12% (i.e., the maximum allowable BAC in the alcohol drinking sessions in this study) or higher at least once in the prior 30 days
* Report at least four days with heavy episodic drinking (i.e., 4 or more drinks for women and 5 or more drinks for men) out of the prior 30 days
* Report having consumed at least one alcoholic drink during a minimum of 12 days out of the prior 30 in order to maximize the likelihood that subjects will choose to drink during the self-administration portion of the laboratory sessions.
* Meet, at minimum, DSM-5 criteria for a mild alcohol use disorder (i.e., meet at least 2 diagnostic criteria)
* Perform within 2 standard deviations of normative levels both with regard to reaction time and number of errors on the cued go/no-go task at in-person screening
* Have an iphone/iOS-compatible phone that they are willing to use for study-related tasks (field use-only participants from outside of the Gainesville area, only; local participants will have an opportunity to borrow a study phone)

Exclusion Criteria:

* Be seeking treatment for alcohol or other addictive behaviors or have been in inpatient or intensive outpatient treatment within the past 12 months
* Have used a smartphone application to facilitate moderate drinking more than 1 time within the past 12 months
* Provide two positive breath alcohol concentration (BrAC) readings (i.e., > 0.00%) at an in-person screening appointment or on the day of the alcohol drinking session. After participants blow their first positive BrAC, they will be allowed to reschedule and participate at another time, however if they blow a second positive BrAC, they will be excluded from this study and offered referrals for alcohol treatment.
* Have positive urine screen results at the in-person screening or on the day of an alcohol drinking session for opiates, cocaine, phencyclidine, amphetamines, methamphetamine, barbiturates, methadone or benzodiazepines.
* Meet criteria for current nicotine dependence or dependence on any other drug, excluding alcohol.
* Report current use of psychotropic drugs including anxiolytics and antidepressants.
* Have received a prescription for any psychotropic drug in the 30 days prior to study enrollment
* Be psychotic or otherwise severely psychiatrically disabled
* Report a history of a medical condition that would contraindicate the consumption of alcohol (e.g., liver disease, cardiac abnormality, pancreatitis, diabetes, neurological problems, and gastrointestinal disorders).
* Have a history of clinically significant withdrawal from alcohol, defined as any one of the following: a) a lifetime history of seizures, delirium, or hallucinations during alcohol withdrawal; b) a Clinical Institute Withdrawal Assessment scale (CIWA-Ar, Sullivan et al., 1989) score > 8; c) a report of drinking to avoid withdrawal symptoms in the past 12 months; or d) a lifetime history of medical treatment for withdrawal.
* A woman who is pregnant, nursing, or refuses to use a reliable method of birth control.
* Report disliking vodka or vodka mixed drinks. Vodka is the alcoholic beverage participants to be used in the proposed study
* Body weight less than 110 pounds or greater than 220 pounds
* Be colorblind
* Be a Foreign National

Ages: 21 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2024-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Liana Hone, MS, MPH, PHD, Principal Investigator — University of Florida
Locations (1):
- UF Health at the University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Control App Condition: Young Adult Drinkers will be randomized to 1 of the 3 app conditions (Control App Version; Standard App Version; Experimental, Feedback App Version). The apps will be tested both during a laboratory alcohol drinking session and a 4-week period outside the lab in which they can use this technology in actual drinking situations. For the 4-week period outside the lab, all participants will use the experimental app for 2 weeks in real drinking occasions and not use it the other 2 weeks.
  Control App Version: The control version is a smartphone-compatible CGNG. The cued go/no-go (CGNG) tests ability to respond fast to "go" targets (activation) while withholding response to "no-go" targets (inhibition).
- Standard App Condition: Young Adult Drinkers will be randomized to 1 of the 3 app conditions (Control App Version; Standard App Version; Experimental, Feedback App Version). The apps will be tested both during a laboratory alcohol drinking session and a 4-week period outside the lab in which they can use this technology in actual drinking situations. For the 4-week period outside the lab, all participants will use the experimental app for 2 weeks in real drinking occasions and not use it the other 2 weeks.
  Standard App Version: The standard version is the same as the control version with the exception that information about performance (correct or incorrect) is displayed along with RT in ms for a correct response during each inter-trial interval.
- Experimental, Feedback App Condition: Young Adult Drinkers will be randomized to 1 of the 3 app conditions (Control App Version; Standard App Version; Experimental, Feedback App Version). The apps will be tested both during a laboratory alcohol drinking session and a 4-week period outside the lab in which they can use this technology in actual drinking situations. For the 4-week period outside the lab, all participants will use the experimental app for 2 weeks in real drinking occasions and not use it the other 2 weeks.
  Experimental, Feedback App Version: The experimental, feedback version includes the standard plus feedback on RT and inhibition errors compared to pre-drinking. The app will state that there are simple alternatives with invitation to press a box to view advice, based on research that risk information may increase risky behavior if convenient options are not given73. Feedback will be worded non-judgmentally per motivational interviewing tenets.
- Field Period Only Participants: A subset of participants were enrolled to participate in the four-week field period only with no laboratory alcohol drinking session.
Period: Overall Study
Arm/Group | Control App Condition | Standard App Condition | Experimental, Feedback App Condition | Field Period Only Participants
Started | 14 | 12 | 14 | 13
Completed | 13 | 12 | 14 | 13
Not Completed | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control App Group | Standard App Group | Experimental, Feedback App Group | Field Period Only Participants | Total
Number analyzed (Participants) | 14 | 12 | 14 | 13 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 12 | 14 | 13 | 53
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.07 (1.44) | 22.08 (1.08) | 22.07 (1.49) | 21.69 (0.95) | 21.98 (1.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 3 | 10 | 28
  Male | 5 | 6 | 11 | 3 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 4 | 1 | 14
  Not Hispanic or Latino | 9 | 8 | 10 | 12 | 39
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 1 | 1 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 13 | 9 | 13 | 12 | 47
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 14 | 12 | 14 | 13 | 53
intensity on State Version of the Alcohol Purchase Task [Mean (Standard Deviation); unit: drinks] — The State Version of the Alcohol Purchase Task is a behavioral economic measure capturing number of drinks participants report an intention to consume now at different price points, provided they were able to drink. Hypothetical costs range from free to $15 each. Higher numbers of self-reported, intended drinks indicates greater motivation to consume alcohol. At each price point, number of drinks can range from 0 to 25. The Alcohol Purchase Task yields several variables, but in this outcome, we considered only intensity, i.e., number of drinks one reports they would have if they were free.
  drinks | 6.92 (3.28) | 7.33 (3.63) | 6.71 (4.48) | 6.97 (3.76) | 6.97 (3.76)
drinks per drinking day [Mean (Standard Deviation); unit: standard alcoholic drinks] | 5.28 (1.28) | 6.27 (3.04) | 5.04 (0.99) | 5.47 (1.38) | 5.49 (1.81)

OUTCOME MEASURES:

1. Primary Outcome: Number of Alcoholic Drinks Intended to Consume if They Were Free (i.e., Intensity)
Description: Number of alcoholic drinks participants report an intention to consume at no cost on the state version of the Alcohol Purchase Task following alcohol administration in the lab. The State Version of the Alcohol Purchase Task is a behavioral economic measure capturing number of drinks participants report an intention to consume now at different price points, provided they were able to drink. Hypothetical costs range from free to $15 each. Higher numbers of self-reported, intended drinks indicates greater motivation to consume alcohol. At each price point, number of drinks can range from 0 to 25. The Alcohol Purchase Task yields several variables, but in this outcome, we considered only intensity, i.e., number of drinks one reports they would have if they were free.
Time Frame: Day 1
Population: Only participants who completed a laboratory alcohol administration session
Measure: Mean (Standard Deviation); unit: drinks
Arm/Group | Control App Group | Standard App Group | Experimental, Feedback App Group
Number analyzed (Participants) | 13 | 12 | 14
drinks | 6.92 (3.28) | 7.33 (3.63) | 6.71 (4.48)
Statistical Analysis 1: Comparison: Control App Group vs Standard App Group vs Experimental, Feedback App Group; Test type: Superiority; p = 0.97, ANOVA

2. Primary Outcome: Change in Number of Alcoholic Drinks Consumed Per Occasion
Description: Entails comparisons of alcoholic drinks consumed per occasion between the 2 weeks participants had full app access vs. the 2 weeks they did not have full app access during the 4-week field use period after the alcohol drinking session.
Time Frame: Two weeks with full app access versus two weeks without during the 4-week field use period
Population: The 4-arm approach was appropriate for Primary Aim 1 when participants were randomized to 1 of 3 experimental conditions in the lab, as opposed to those who did not complete a lab session. However, for these field use analyses, since all participants had the same experience, within subjects comparisons among the entire sample that completed the field period were most appropriate. Thus, these analyses include those who completed a lab session and those who completed the field use period only
Measure: Mean (Standard Deviation); unit: standard alcoholic drinks
Groups:
- All Participants Who Completed the Field Use Period: This is a single group, within-subjects comparison of number of drinks consumed per occasion during the two weeks when participants had full access to the app with its intervention components versus two weeks when they only completed daily questionnaires using the app and did not have access to the app's intervention components. All participants who completed the field use period were included in these analyses.
Arm/Group | All Participants Who Completed the Field Use Period
Number analyzed (Participants) | 53
standard alcoholic drinks
  2 weeks with full intervention app access | 5.37 (2.60)
  2 weeks without full intervention app access | 5.01 (2.31)
Statistical Analysis 1: Comparison: All Participants Who Completed the Field Use Period; Within subjects comparison of drinks per drinking day with full intervention app access versus daily assessment via the app only; Test type: Superiority; p = .232, t-test, 2 sided; Mean Difference (Final Values) = 0.36, 95% CI 2-sided [-0.24 to 0.95], Standard Deviation 2.09

ADVERSE EVENTS:
Time Frame: A period up to about six weeks including screening period, laboratory session and field use period.
Description: standard adverse event and serious adverse event descriptions were used
Groups:
- Experimental, Feedback App During Field Use Period: Participants enrolled to participate in the four-week field period with or without the laboratory alcohol drinking session.
Arm/Group | Control App Condition | Standard App Condition | Experimental, Feedback App Condition | Experimental, Feedback App During Field Use Period
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/12 | 0/14 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/12 | 0/14 | 0/53
Other Adverse Events (participants affected / at risk) | 0/14 | 0/12 | 0/14 | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-28): https://cdn.clinicaltrials.gov/large-docs/59/NCT04243759/Prot_SAP_000.pdf
  • Informed Consent Form (2023-07-12): https://cdn.clinicaltrials.gov/large-docs/59/NCT04243759/ICF_001.pdf